CLINICAL TRIAL: NCT01938664
Title: Pilot Study of Candesartan: An Angiotensin Receptor Blocker as a Treatment for Cocaine Dependence
Brief Title: A Pilot Study of Candesartan as a Treatment for Cocaine Dependence
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Results of interim efficacy analysis showed results were not promising.
Sponsor: Baylor College of Medicine (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Thomas R. Kosten, MD, Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H-32241; 5P50DA018197-09 (NIH)
Record Dates: First submitted 2013-09-05; First posted 2013-09-10 (Estimated); Results first posted 2019-08-26 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-08

CONDITIONS: Cocaine Dependence
Keywords: cocaine; dependence; pharmacotherapy
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — candesartan; candesartan cilexetil

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Candesartan w Cognitive Behavior Therapy (Experimental): Titration up to 8mg through week 1. Continue on 8mg thru wk 8. CBT optional thru study.
  Interventions: Drug: Candesartan with CBT
- Placebo w Cognitive Behavior Therapy (Placebo Comparator): Sugar pill to mimic Candesartan for study duration. CBT optional thru study.
  Interventions: Other: Placebo with CBT

INTERVENTIONS:
Drug: Candesartan with CBT — 8 mg, po (by mouth)
  Other Names: atacand
  Arms: Candesartan w Cognitive Behavior Therapy
Other: Placebo with CBT
  Arms: Placebo w Cognitive Behavior Therapy

SUMMARY:
The purpose of this study is to see if a drug called Candesartan will help to reduce use of cocaine.

DETAILED DESCRIPTION:
The noradrenergic system may play an important role in cocaine addiction in humans. Angiotensin II (Ang II) is known to enhance noradrenergic activity, which contributes to effects on blood pressure and sympathetic nervous system responses to stress. Inhibition of Ang II has been shown to reduce cravings for stimulants, including cocaine and methamphetamine.

This clinical trial among 75 cocaine-dependent subjects is designed to test the efficacy of the Angiotensin II receptor antagonist, Candesartan, for treatment of cocaine dependence. The results of this study will provide medical safety and efficacy data, and will guide future pharmacotherapy trials using this class of medications for cocaine addiction.

This 8-week trial includes a 1-week titration of the medication and 7-weeks of full dose medication (weeks 2-8), with all subjects receiving the active agent.

At the conclusion of the trial, subjects who wish to be referred to an appropriate treatment program or treatment research program will be assisted with a referral.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for study entry, all subjects must satisfy the following criteria:

1. Age 18 to 64 years inclusive;
2. Females either must be of non-child bearing potential (i.e., surgically sterilized or postmenopausal) or must be using adequate contraception, have a negative pregnancy test, and must agree to continue to use such precautions for the duration of the study.
3. Meets Diagnostic and Statistical Manual of Mental Disorders Fourth Edition (DSM-IV-TR) criteria for a principal diagnosis of cocaine dependence as confirmed by the MINI and/or as per PI/study investigator's examination of the patient during screening. (Per DSM-IV-TR, principal diagnosis is the condition that is the primary target of treatment at the time of presentation);
4. Motivated to discontinue or reduce cocaine use during the period of the study, as evidenced both by the judgment of the Investigator or designee and by the subject's compliance level with the requirement for attendance at clinic visits such that the urine sample requirements for inclusion criteria #6 is fully met;
5. Has a positive pattern of cocaine usage as determined by provision of at least one cocaine positive urine sample (benzoylecgonine (BE) level at least 300 ng/ml) during the screening period; typically conducted over a 7-14 day period.
6. In good general health as determined by self-reported and/or computer-based medical history, general clinical examination, and laboratory tests;
7. Has provided written informed consent.
8. Are cooperative, willing and able to participate and adhere to the protocol requirements

Exclusion Criteria:

Subjects will be excluded from the study if one or more of the following statements are applicable:

1. Subject is taking angiotensin-converting enzyme (ACE) inhibitors such as benazepril (Lotensin, in Lotrel), captopril (Capoten, in Capozide), enalapril (Vasotec, in Lexxel, in Vaseretic), fosinopril (Monopril), lisinopril (Prinivil, Zestril, in Prinzide, in Zestoretic), moexipril (Univasc, in Uniretic), perindopril, (Aceon), quinapril (Accupril, in Accuretic, in Quinaretic), ramipril (Altace), and trandolapril (Mavik, in Tarka); lithium (Eskalith Controlled-Release, Eskalith, Lithobid);
2. Subject is on psychotropic medications, an MAOI, or an opiate antagonist;
3. Subject is currently taking a dopaminergic, dopamine-blocking, dopamine-modulating, or other central dopamine-altering drug (e.g., antipsychotic drugs); a monoamine oxidase inhibitor (MAOI); or an opiate antagonist;
4. Subject has an unstable medical, neurologic, or psychiatric illness that would interfere with the subject's safety, ability to participate in the study, or the interpretability of data. Subjects who meet the DSM-IV-R criteria for psychosis, schizophrenia, bipolar disorder or clinically significant suicidal ideation as assessed by the PI/study investigator and/or the MINI will be excluded. Subjects who have been taking stable doses of antidepressants for at least 3 months at the time the consent is signed will be allowed onto the study unless those antidepressants are of the types specified under exclusion criteria #3,above;
5. Subject is dependent on benzodiazepines, barbiturates, amphetamines, opiates (including methadone or buprenorphine maintenance treatment) according to the DSM-IV-R and as assessed by the PI/study investigator and/or the MINI; 6
6. Subject is, in the investigator's opinion, at risk of requiring medical detoxification for alcohol dependence during the study;
7. Subject has participated in another clinical trial or received any other investigational compound within 7 days prior to being randomized into this study;
8. Significant medical conditions (e.g., major cardiovascular, renal, endocrine, hepatic disorders, immunosuppressive disorders) such as abnormal liver function (with laboratory findings of serum glutamic oxaloacetic transaminase (SGOT) or serum glutamic-pyruvic transaminase (SGPT) greater than three times normal), hypotension, hypertension, a current cardiac condition, and those having a high risk of cardiovascular disease, seizure disorder, or another significant underlying medical condition which would contraindicate Candesartan treatment;
9. Upon review of a compilation of screening data, at the discretion of the PI/study investigator, a participant may be excluded from the study if they test positive during the screening process for any substance other than cocaine or marijuana;
10. Female subjects with a positive pregnancy test, lactating mothers, women refusing to agree to pregnancy tests during the study, women who are planning to become pregnant during the period of the trial or women of child-bearing potential who refuse to agree to use adequate contraception during the study. Acceptable contraceptive methods are oral or parenteral hormonal contraceptives, intrauterine device (IUD), or barrier and spermicide, but not abstinence; OR Male subjects refusing to agree to use adequate contraception during the study, or males who are part of a couple planning to become pregnant during the period of the trial;
11. Any other factor that per the Investigator/designee would make the subject unsafe or unsuitable for the study.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2013-01; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Kosten, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Michael E. DeBakey VA Medical Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo w Cognitive Behavior Therapy: Sugar pill to mimic Candesartan for study duration. CBT optional thru study.
  Placebo with CBT
Period: Overall Study
Arm/Group | Candesartan w Cognitive Behavior Therapy | Placebo w Cognitive Behavior Therapy
Started | 20 | 10
Completed (This only includes subjects that completed 4 weeks of study treatment until the efficacy analysis.) | 5 | 0
Not Completed | 15 | 10

BASELINE CHARACTERISTICS:
Groups:
- Candesartan w Cognitive Behavior Therapy: Titration up to 8mg wk 1-4. Continue on 8mg thru wk 8. CBT optional thru study.
  Candesartan with CBT: 8 mg, po (by mouth)
- Total: Total of all reporting groups
Arm/Group | Candesartan w Cognitive Behavior Therapy | Placebo w Cognitive Behavior Therapy | Total
Number analyzed (Participants) | 20 | 10 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 10 | 30
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 20 | 10 | 30

OUTCOME MEASURES:

1. Primary Outcome: # of Participants With Presence of Cocaine Metabolites Via Urinalysis
Time Frame: thrice weekly, baseline thru week 8
Measure: Number; unit: participants
Arm/Group | Candesartan w Cognitive Behavior Therapy | Placebo w Cognitive Behavior Therapy
Number analyzed (Participants) | 20 | 10
participants | 20 | 10

2. Secondary Outcome: # of Participants Retained in Study
Time Frame: 8 weeks
Measure: Number; unit: participants
Arm/Group | Candesartan w Cognitive Behavior Therapy | Placebo w Cognitive Behavior Therapy
Number analyzed (Participants) | 20 | 10
participants | 5 | 0

3. Secondary Outcome: # of Participants With Adverse Events
Description: Candesartan will be well tolerated without significant side effects.
Time Frame: 8 weeks
Measure: Number; unit: participants
Arm/Group | Candesartan w Cognitive Behavior Therapy | Placebo w Cognitive Behavior Therapy
Number analyzed (Participants) | 20 | 10
participants | 0 | 0

ADVERSE EVENTS:
Arm/Group | Candesartan w Cognitive Behavior Therapy | Placebo w Cognitive Behavior Therapy
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/10
Other Adverse Events (participants affected / at risk) | 0/20 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No